CLINICAL TRIAL: NCT03928171
Title: The Effect of Intra-abdominal Pressure on Peritoneal Perfusion During Laparoscopic Colorectal Surgery: a Pilot Study
Brief Title: The Effect of Intra-abdominal Pressure on Peritoneal Perfusion During Laparoscopic Colorectal Surgery
Acronym: PERFUSION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2018-4313
Record Dates: First submitted 2019-04-23; First posted 2019-04-26 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2019-04

CONDITIONS: Laparoscopic Surgery; Pneumoperitoneum
Keywords: Laparoscopic surgery; Pneumoperitoneum; Peritoneal perfusion; Intra-abdominal pressure
MeSH Terms: conditions — Pneumoperitoneum

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intra-abdominal pressure of 8 mmHg (Experimental): The laparoscopy insufflator is set to a pressure of 8 mmHg
  Interventions: Other: Intra-abdominal pressure during laparoscopy
- Intra-abdominal pressure of 12 mmHg (Experimental): The laparoscopy insufflator is set to a pressure of 12 mmHg
  Interventions: Other: Intra-abdominal pressure during laparoscopy
- Intra-abdominal pressure of 16 mmHg (Experimental): The laparoscopy insufflator is set to a pressure of 16 mmHg
  Interventions: Other: Intra-abdominal pressure during laparoscopy

INTERVENTIONS:
Other: Intra-abdominal pressure during laparoscopy — Insufflation pressure of the abdomen during laparoscopy

SUMMARY:
Peritoneal perfusion during laparoscopic surgery is quantified by video recording after intravenous injection of indocyanine green at a pneumoperitoneum pressure of 8, 12 and 16 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥ 18 years old)
* Scheduled for robot-assisted colorectal laparoscopic surgery

Exclusion Criteria:

* Severe liver- or renal disease
* Pregnancy or lactation
* Planned diagnostics or treatment with radioactive iodine < 1 week after surgery
* BMI >35 kg/m2
* Known or suspected hypersensitivity to indocyanine green, sodium iodide or iodine
* Hyperthyroidism or thyroid adenomas
* Use of medication interfering with ICG absorption as listed in the summary of product characteristics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2018-12-24 (Actual)

PRIMARY OUTCOMES:
Peritoneal perfusion | 3 minutes after intravenous injection of indocyanine green
  Perfusion is quantified by video recording of the parietal peritoneum using the Firefly fluorescence module of the DaVinci surgical robot after intravenous injection of 0.2mg/kg indocyanine green. Fluorescent intensity in [-] over time is plotted in MATLAB, maximum fluorescent intensity and time to reach maximum fluorescent intensity are extracted.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel C Warlé, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Albers KI, Polat F, Loonen T, Graat LJ, Mulier JP, Snoeck MM, Panhuizen IF, Vermulst AA, Scheffer GJ, Warle MC. Visualising improved peritoneal perfusion at lower intra-abdominal pressure by fluorescent imaging during laparoscopic surgery: A randomised controlled study. Int J Surg. 2020 May;77:8-13. doi: 10.1016/j.ijsu.2020.03.019. Epub 2020 Mar 17. PMID 32194255